CLINICAL TRIAL: NCT01575704
Title: Physical Exercise Therapy in Pediatric Stem Cell Transplantation (BISON- Bewegungstherapie in Der Pädiatrischen Stammzelltransplantation)
Brief Title: Physical Exercise Therapy in Pediatric Stem Cell Transplantation
Acronym: BISON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Institut für Sportwissenschaften, Frankfurt (Unknown); Fresenius University of Applied Science (Other)
Responsible Party: Principal Investigator, Peter Bader, Head Department of Stem Cell Transplantation and Immunology, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BISON01042011
Record Dates: First submitted 2012-03-08; First posted 2012-04-11 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Hematopoetic Stem Cell Transplantation
Keywords: Exercise; Hematopoetic cell transplantation; Children
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sport (Experimental)
  Interventions: Other: Exercise
- Control (Other)
  Interventions: Other: Mental Training

INTERVENTIONS:
Other: Exercise — Supervised exercise training (aerobic, resistance, flexibility), 5 times per week
  Arms: Sport
Other: Mental Training — Memorial/ mental training and relaxation, 5 times per week
  Arms: Control

SUMMARY:
The purpose of this randomized controlled two-part study examines the effects of a structured sports intervention before, during and after hematopoetic stem cell transplantation (hsct) in children and adolescents.

The main aspects in the sports groups are resistance, endurance and flexibility training. The control group performs a mental training as well as relaxation exercises.

ELIGIBILITY:
Inclusion Criteria:

* Indication for hsct
* Informed consent signed

Exclusion Criteria:

* Contraindication for exercise
* Age < 5 years
* Insuperable language barrier
* Orthopeadical, cardiological or neurological indication for physical therapy

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Muscle strength | change between hospital admission and discharge (approximately 4-6 weeks) and 3 months and 6 months after transplantation
  Upper limb: hand grip strength with JAMAR dynamometry; Lower limb: maximal isometric voluntary strength of M. quadriceps femoris

SECONDARY OUTCOMES:
Fatigue | change between hospital admission and discharge (approximately 4-6 weeks) and 3 months and 6 months after transplantation
  Pediatric Quality of Life Inventory (PedsQL)
Biomarker in blood | daily
  Hematological and immunological reconstitution
Body composition | one time per week and change between 3 months and 6 months after transplantation
  Bioelectrical Impedance Analyse (BIA; Data Input GmbH)
Endurance performance | change between hospital admission and discharge (approximately 4-6 weeks) and 3 months and 6 months after transplantation
  6-Minute-Walking-Test (6MWT); Ergospirometry and Echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Senn-Malashonak A, Wallek S, Schmidt K, Rosenhagen A, Vogt L, Bader P, Banzer W. Psychophysical effects of an exercise therapy during pediatric stem cell transplantation: a randomized controlled trial. Bone Marrow Transplant. 2019 Nov;54(11):1827-1835. doi: 10.1038/s41409-019-0535-z. Epub 2019 May 14. PMID 31089282